CLINICAL TRIAL: NCT02581202
Title: ProSpective, MultI-Center, Observational PrograM to Assess the Effectiveness of Dual TheraPy (Lopinavir/Ritonavir + LamivudinE) in Treatment-Experienced HIV Infected Patients in the Routine Clinical Settings of the Russian Federation (SIMPLE)
Brief Title: The Effectiveness of Dual Therapy (Lopinavir/Ritonavir + LamivudinE) in Treatment-Experienced HIV Infected Patients in the Russian Federation
Acronym: SIMPLE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-452
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2018-05

CONDITIONS: HIV-1 Infection
Keywords: antiretroviral therapy
MeSH Terms: interventions — Lopinavir; Lamivudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-1 infected participants: HIV-1-infected participants on any triple highly active antiretroviral therapy (HAART) with plasma HIV-1 ribonucleic acid (RNA) level < 50 copies/mL for at least 6 months (two consequently plasma HIV-1 RNA levels) transferred as medically appropriate to lopinavir with ritonavir plus lamivudine (LPV/r+3TC) as decided by the physician in the routine clinical settings. Or HIV-1 infected participants who were switched on the dual therapy (LPV/r+3TC) no more than 60 days prior to enrollment.
  Interventions: Drug: lopinavir/ritonavir; Drug: lamivudine

INTERVENTIONS:
Drug: lopinavir/ritonavir — tablet
Drug: lamivudine — tablet

SUMMARY:
This study seeks to assess the virologic effectiveness of dual therapy (lopinavir/ ritonavir (LPV/r) + lamivudine (3TC)) in treatment-experienced human immunodeficiency virus 1 (HIV-1) infected participants with an undetectable plasma HIV-1 (ribonucleic acid) RNA level (for at least 6 months) at the 48 week time point of treatment in the routine clinical settings of the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older (male and female).
2. HIV-1 infected patients on any triple HAART with plasma HIV-1 RNA level <50 copies/mL for at least 6 months (two consequently plasma HIV-1 RNA levels) transferred as medically appropriate to LPV/r + 3TC as decided by the physician in the routine clinical settings. Or HIV-1 infected patients who were switched on the dual therapy (LPV/r + 3TC) no more than 60 days ago.
3. Cumulative HAART experience at least 6 months.
4. Authorization (Consent) for Use/Disclosure of Data signed by the patient.

Exclusion Criteria:

1. Contraindications to lopinavir/ritonavir and lamivudine
2. Previous participation in this program

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected participants on any triple HAART with undetectable plasma HIV-1 RNA level for at least 6 months (two consequently plasma HIV-1 RNA levels) transferred as medically appropriate to LPV/r + 3TC in the routine clinical settings.
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2015-12-21; Primary Completion 2017-05-27 (Actual); Study Completion 2017-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Strugovschikov, MD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Immunodeficiency Virus 1 (HIV-1) Infected Participants: HIV-1-infected participants on any triple highly active antiretroviral therapy (HAART) with plasma HIV-1 ribonucleic acid (RNA) level < 50 copies/mL for at least 6 months (two consequently plasma HIV-1 RNA levels) transferred as medically appropriate to lopinavir with ritonavir plus lamivudine (LPV/r+3TC) as decided by the physician in the routine clinical settings. Or HIV-1 infected participants who were switched on the dual therapy (LPV/r+3TC) no more than 60 days prior to enrollment.
Period: Overall Study
Arm/Group | Human Immunodeficiency Virus 1 (HIV-1) Infected Participants
Started | 216
Completed | 202
Not Completed | 14
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 5
Not completed — Pregnancy | 3

BASELINE CHARACTERISTICS:
Groups:
- HIV-1 Infected Participants: HIV-1infected participants on any triple HAART with plasma HIV-1 RNA level < 50 copies/mL for at least 6 months (two consequently plasma HIV-1 RNA levels) transferred as medically appropriate to LPV/r+3TC as decided by the physician in the routine clinical settings. Or HIV-1 infected participants who were switched on the dual therapy (LPV/r+3TC) no more than 60 days prior to enrollment.
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144
  Male | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 216
Absolute HIV-1 RNA Viral Load (Untransformed Data) [Mean (Standard Deviation); unit: copies/mL] — Statistics for absolute HIV-1 RNA viral load, where all participants with undetectable HIV-1-RNA viral load data were included into calculations with half of the lower indication limit (50/2 copies/mL, or 25.00 copies/mL).
  copies/mL | 25.00 (0.000)
HIV-1 RNA Viral Load (Log10-Transformed Data) [Mean (Standard Deviation); unit: log10 copies/mL] | 3.22 (0.000)
CD4+T-Cell Counts (%) [Mean (Standard Deviation); unit: percentage of lymphocytes that are CD4+] | 31.44 (8.396)
CD4+T-Cell Counts (cells/mm^3) [Mean (Standard Deviation); unit: cells/mm^3] | 641.37 (251.417)
Arm Circumference [Mean (Standard Deviation); unit: cm] | 30.03 (5.290)
Hip Circumference [Mean (Standard Deviation); unit: cm] | 53.92 (7.096)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 82.79 (11.579)
Alanine Aminotransferase (U/L) [Mean (Standard Deviation); unit: U/L] — Population: participants with an evaluable baseline assessment
  U/L
    number analyzed (Participants) | 200
    (all) | 31.48 (33.910)
Alanine Aminotransferase (µmol/L) [Mean (Standard Deviation); unit: µmol/L] — Population: participants with an evaluable baseline assessment
  µmol/L
    number analyzed (Participants) | 16
    (all) | 20.75 (7.979)
Aspartate Aminotransferase (U/L) [Mean (Standard Deviation); unit: U/L] — Population: participants with an evaluable baseline assessment
  U/L
    number analyzed (Participants) | 200
    (all) | 27.69 (22.913)
Aspartate Aminotransferase (µmol/L) [Mean (Standard Deviation); unit: µmol/L] — Population: participants with an evaluable baseline assessment
  µmol/L
    number analyzed (Participants) | 16
    (all) | 21.56 (11.933)
Glucose [Mean (Standard Deviation); unit: mmol/L] | 4.96 (0.590)
High Density Lipoprotein (HDL) [Mean (Standard Deviation); unit: mmol/L] — Population: participants with an evaluable baseline assessment
  mmol/L
    number analyzed (Participants) | 117
    (all) | 1.45 (0.479)
Insulin [Mean (Standard Deviation); unit: µEq/mL] — Population: participants with an evaluable baseline assessment
  µEq/mL
    number analyzed (Participants) | 35
    (all) | 9.32 (2.085)
Low Density Lipoprotein (LDL) [Mean (Standard Deviation); unit: mmol/L] — Population: participants with an evaluable baseline assessment
  mmol/L
    number analyzed (Participants) | 106
    (all) | 2.75 (0.866)
Serum Creatinine [Mean (Standard Deviation); unit: µmol/L] — Population: participants with an evaluable baseline assessment
  µmol/L
    number analyzed (Participants) | 208
    (all) | 78.61 (18.136)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] — Population: participants with an evaluable baseline assessment
  mmol/L
    number analyzed (Participants) | 214
    (all) | 5.04 (0.980)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] — Population: participants with an evaluable assessment at baseline
  mmol/L
    number analyzed (Participants) | 189
    (all) | 2.29 (8.107)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on Dual Therapy (LPV/r + 3TC) With Undetectable HIV-1 RNA Level at Week 48
Time Frame: Week 48
Population: Participants with an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HIV-1 Infected Participants: HIV-1infected patients on any triple HAART with plasma HIV-1 RNA level < 50 copies/mL for at least 6 months (two consequently plasma HIV-1 RNA levels) transferred as medically appropriate to LPV/r+3TC as decided by the physician in the routine clinical settings. Or HIV-1 infected patients who were switched on the dual therapy (LPV/r+3TC) no more than 60 days prior to enrollment.
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 201
percentage of participants | 100 [98.18 to 100.0]

2. Secondary Outcome: Percentage of Participants on Dual Therapy (LPV/r + 3TC) With Undetectable HIV-1 RNA Level at Week 24
Time Frame: Week 24
Population: Participants with an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 203
percentage of participants | 99.5 [97.29 to 99.99]

3. Secondary Outcome: Absolute Values and Change From Baseline (BL) in HIV-1- RNA Viral Load at Week 24 (Untransformed Data)
Time Frame: Baseline, Week 24
Population: Participants with data on HIV-1 RNA viral load at given time point.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 203
copies/mL
  Absolute values | 25.22 (3.158)
  Change from BL | 0.22 (3.158)

4. Secondary Outcome: Absolute Values and Change From Baseline (BL) in HIV-1- RNA Viral Load at Week 24 (Base-10 Logarithm Transformed Data)
Time Frame: Baseline, Week 24
Population: Participants with data on HIV-1 RNA viral load at given time point.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 203
log10 copies/mL
  Absolute values | 3.22 (0.072)
  Change from BL | 0.01 (0.072)

5. Secondary Outcome: Absolute Values and Change From Baseline in HIV-1- RNA Viral Load at Week 48 (Untransformed Data)
Description: Statistics for absolute HIV-1 RNA viral load, where all participants with undetectable HIV-1-RNA viral load data were included into calculations with half of the lower indication limit (50/2 copies/mL, or 25.00 copies/mL).
Time Frame: Baseline, Week 48
Population: Participants with data on HIV-1 RNA viral load at given time point.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 201
copies/mL
  Absolute values | 25.00 (0.000)
  Change from BL | 0.00 (0.000)

6. Secondary Outcome: Absolute Values and Change From Baseline in HIV-1- RNA Viral Load at Week 48 (Base-10 Logarithm Transformed Data)
Time Frame: Baseline, Week 48
Population: Participants with data on HIV-1 RNA viral load at given time point.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 201
log10 copies/mL
  Absolute values | 3.22 (0.000)
  Change from BL | 0.000 (0.000)

7. Secondary Outcome: Absolute Values and Change From Baseline in CD4+ T-cell Counts (%) at Week 24
Time Frame: Baseline, Week 24
Population: Participants with valid measurements at given time point.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes that are CD4+
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 205
percentage of lymphocytes that are CD4+
  Absolute values | 32.50 (7.554)
  Change from BL | 0.96 (4.879)

8. Secondary Outcome: Absolute Values and Change From Baseline in CD4+ T-cell Counts (%) at Week 48
Time Frame: Baseline, Week 48
Population: Participants with valid measurements at given time point.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes that are CD4+
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 202
percentage of lymphocytes that are CD4+
  Absolute values | 33.11 (7.860)
  Change from BL | 1.43 (6.314)

9. Secondary Outcome: Absolute Values and Change From Baseline in CD4+ T-cell Counts (Cells/mm^3) at Week 24
Time Frame: Baseline, Week 24
Population: Participants with valid measurements at given time point.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 205
cells/mm^3
  Absolute values | 703.43 (223.790)
  Change from BL | 64.70 (165.060)

10. Secondary Outcome: Absolute Values and Change From Baseline in CD4+ T-cell Counts (Cells/mm^3) at Week 48
Time Frame: Baseline, Week 48
Population: Participants with valid measurements at given time point.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 202
cells/mm^3
  Absolute values | 752.44 (234.366)
  Change from BL | 111.75 (184.477)

11. Secondary Outcome: Number of Participants Who Developed Resistance to Nucleoside Reverse Transcriptase Inhibitors (NRTIs), Non-nucleoside Reverse Transcriptase Inhibitors (NNRTIs), and Protease Inhibitors (PIs)
Time Frame: Week 48
Population: Participants with HIV-1 RNA viral load detected levels of ≥ 50 copies/mL up to Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 5
Participants
  NRTI | 1
  NNRTI | 1
  PI | 0

12. Secondary Outcome: Absolute Values and Change From Baseline in Anthropometric Measurements At Week 24
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 205
cm
  Absolute values: arm circumference | 29.82 (4.617)
  Change from BL: arm circumference | -0.38 (2.953)
  Absolute values: hip circumference | 54.62 (8.112)
  Change from BL: hip circumference | 0.57 (5.575)
  Absolute values: waist circumference | 83.29 (12.282)
  Change from BL: waist circumference | 0.31 (5.998)

13. Secondary Outcome: Absolute Values and Change From Baseline in Anthropometric Measurements At Week 48
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 202
cm
  Absolute values: arm circumference | 30.05 (4.781)
  Change from BL: arm circumference | -0.20 (2.935)
  Absolute values: hip circumference | 55.25 (8.395)
  Change from BL: hip circumference | 1.14 (6.739)
  Absolute values: waist circumference | 83.64 (12.742)
  Change from BL: waist circumference | 0.63 (6.026)

14. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Alanine Aminotransferase (U/L)
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 188
U/L
  Absolute values | 29.37 (28.674)
  Change from BL | -1.31 (21.483)

15. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Alanine Aminotransferase (U/L)
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 186
U/L
  Absolute values | 28.35 (28.386)
  Change from BL | -2.14 (25.666)

16. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Alanine Aminotransferase (µmol/L)
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 16
µmol/L
  Absolute values | 39.81 (36.996)
  Change from BL | 19.06 (35.093)

17. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Alanine Aminotransferase (µmol/L)
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 16
µmol/L
  Absolute values | 27.56 (11.950)
  Change from BL | 6.81 (10.950)

18. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Aspartate Aminotransferase (U/L)
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 187
U/L
  Absolute values | 26.90 (21.575)
  Change from BL | -0.38 (17.234)

19. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Aspartate Aminotransferase (U/L)
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 185
U/L
  Absolute values | 26.92 (21.050)
  Change from BL | -0.49 (20.640)

20. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Aspartate Aminotransferase (µmol/L)
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 16
µmol/L
  Absolute values | 46.56 (65.596)
  Change from BL | 25.00 (65.300)

21. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Aspartate Aminotransferase (µmol/L)
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 16
µmol/L
  Absolute values | 27.19 (14.543)
  Change from BL | 5.63 (10.966)

22. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Glucose
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 204
mmol/L
  Absolute values | 4.88 (0.690)
  Change from BL | -0.10 (0.838)

23. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Glucose
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 202
mmol/L
  Absolute values | 4.83 (0.755)
  Change from BL | -0.16 (0.818)

24. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: HDL
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 110
mmol/L
  Absolute values | 1.53 (0.594)
  Change from BL: number analyzed (Participants) | 92
  Change from BL | 0.07 (0.622)

25. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: HDL
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 97
mmol/L
  Absolute values | 1.43 (0.465)
  Change from BL: number analyzed (Participants) | 90
  Change from BL | -0.00 (0.568)

26. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Insulin
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: µEq/mL
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 35
µEq/mL
  Absolute values | 10.00 (2.342)
  Change from BL | 0.68 (2.683)

27. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Insulin
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: µEq/mL
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 33
µEq/mL
  Absolute values | 10.00 (2.358)
  Change from BL | 0.69 (2.760)

28. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: LDL
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 111
mmol/L
  Absolute values | 2.66 (0.902)
  Change from BL: number analyzed (Participants) | 92
  Change from BL | -0.07 (0.726)

29. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: LDL
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 94
mmol/L
  Absolute values | 2.92 (0.874)
  Change from BL: number analyzed (Participants) | 86
  Change from BL | 0.14 (0.893)

30. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Serum Creatinine
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 196
µmol/L
  Absolute values | 81.50 (19.488)
  Change from BL: number analyzed (Participants) | 188
  Change from BL | 2.36 (15.286)

31. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Serum Creatinine
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 184
µmol/L
  Absolute values | 82.13 (19.096)
  Change from BL: number analyzed (Participants) | 176
  Change from BL | 2.75 (15.801)

32. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Total Cholesterol
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 199
mmol/L
  Absolute values | 5.11 (0.951)
  Change from BL: number analyzed (Participants) | 197
  Change from BL | 0.07 (0.928)

33. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Total Cholesterol
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 187
mmol/L
  Absolute values | 5.12 (1.118)
  Change from BL: number analyzed (Participants) | 185
  Change from BL | 0.11 (0.986)

34. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 24: Triglycerides
Time Frame: Baseline, Week 24
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 171
mmol/L
  Absolute values | 1.72 (1.025)
  Change from BL: number analyzed (Participants) | 149
  Change from BL | -0.70 (9.106)

35. Secondary Outcome: Absolute Values and Change From Baseline in Metabolic Parameters at Week 48: Triglycerides
Time Frame: Baseline, Week 48
Population: Participants with measurements at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 159
mmol/L
  Absolute values | 1.61 (0.832)
  Change from BL: number analyzed (Participants) | 142
  Change from BL | -0.06 (1.313)

36. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events were not recorded in a solicited manner as in an interventional trial, but were recorded by spontaneous reporting in line with the requirements described in European Medicines Agency (EMA) Guideline on Good Pharmacovigilance Practices (GVP) module VI and local pharmacovigilance practice of the Russian Federation.
Time Frame: up to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-1 Infected Participants
Number analyzed (Participants) | 216
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to Week 48
Description: This study is non-interventional. Therefore, adverse events were not recorded in a solicited manner as in an interventional trial, but were recorded by spontaneous reporting in line with the requirements described in EMA Guideline on GVP module VI and local pharmacovigilance practice of the Russian Federation.
Groups:
- HIV-1 Infected Participants: Treatment-experienced HIV-1 infected participants with an undetectable plasma HIV-1 RNA level
  lopinavir/ritonavir: tablet
  Lamivudine: tablet
Arm/Group | HIV-1 Infected Participants
All-Cause Mortality (participants affected / at risk) | 0/216
Serious Adverse Events (participants affected / at risk) | 0/216
Other Adverse Events (participants affected / at risk) | 3/216
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-1 Infected Participants (N=216)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Drug ineffective (General disorders) | 2
Transaminases increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT02581202/Prot_SAP_000.pdf